CLINICAL TRIAL: NCT05272384
Title: A Phase 1 Study of Nivolumab in Combination With ASTX727 in B-cell Lymphoma (NHL or HL) With an Expansion Cohort in Relapsed or Refractory Diffuse Large B-Cell Lymphoma (DLBCL) and Hodgkin Lymphoma (HL)
Brief Title: Testing the Combination of Nivolumab and ASTX727 for Relapsed or Refractory B-Cell Lymphoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2022-01799; NCI-2022-01799 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S22-00427; 10508 (Other: Dana-Farber - Harvard Cancer Center LAO); 10508 (Other: CTEP); P01CA229086 (NIH); P30CA016087 (NIH)
Record Dates: First submitted 2022-03-08; First posted 2022-03-09 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-09

CONDITIONS: Recurrent B-Cell Non-Hodgkin Lymphoma; Recurrent Diffuse Large B-Cell Lymphoma; Recurrent Hodgkin Lymphoma; Refractory B-Cell Non-Hodgkin Lymphoma; Refractory Diffuse Large B-Cell Lymphoma; Refractory Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma, Large B-Cell, Diffuse; Hodgkin Disease | interventions — Specimen Handling; decitabine and cedazuridine drug combination; Nivolumab; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (nivolumab, decitabine and cedazuridine) (Experimental): Patients receive decitabine and cedazuridine PO QD on days 1-3 or 1-5 of each cycle and nivolumab IV over 30 minutes on day 15 of each cycle. Treatment repeats every 28 days for 12 cycles in the absence of disease progression or unacceptable toxicity. Patients with CR, PR, or SD after 12 cycles receive decitabine and cedazuridine for an additional 12 months. Patients also undergo PET/CT and collection of blood samples throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Decitabine and Cedazuridine; Biological: Nivolumab; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Decitabine and Cedazuridine — Given PO
  Other Names: ASTX 727; ASTX-727; ASTX727; C-DEC; CDA Inhibitor E7727/Decitabine Combination Agent ASTX727; Cedazuridine/Decitabine Combination Agent ASTX727; Cedazuridine/Decitabine Tablet; DEC-C; Inaqovi; Inqovi
Biological: Nivolumab — Given IV
  Other Names: ABP 206; BCD-263; BMS 936558; BMS-936558; BMS936558; CMAB819; MDX 1106; MDX-1106; MDX1106; NIVO; Nivolumab Biosimilar ABP 206; Nivolumab Biosimilar BCD-263; Nivolumab Biosimilar CMAB819; ONO 4538; ONO-4538; ONO4538; Opdivo
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT

SUMMARY:
This phase I trial tests the safety, side effects, and best dose of nivolumab in combination with ASTX727 in treating B-cell lymphoma that has come back (relapsed) or does not respond to treatment (refractory). Immunotherapy with monoclonal antibodies, such as nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. ASTX727 consists of the combination of decitabine and cedazuridine. Cedazuridine is in a class of medications called cytidine deaminase inhibitors. It prevents the breakdown of decitabine, making it more available in the body so that decitabine will have a greater effect. Decitabine is in a class of medications called hypomethylation agents. It works by helping the bone marrow produce normal blood cells and by killing abnormal cells in the bone marrow. Giving nivolumab in combination with ASTX727 may shrink and stabilize cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the safety and tolerability of the combination of oral deoxyribonucleic acid (DNA) methyltransferase (DNMT) inhibition and checkpoint inhibition in relapsed or refractory B cell lymphoma (dose escalation) and diffuse large B-cell lymphoma (DLBCL) (dose expansion) or Hodgkin lymphoma (dose expansion).

SECONDARY OBJECTIVES:

I. To observe and record anti-tumor activity. II. To evaluate the response rate (overall response [ORR], complete response [CR], and partial response [PR]), and the progression free survival (PFS) and overall survival (OS) in patients with relapsed or refractory DLBCL treated with the combination of oral DNMT inhibition and checkpoint inhibition.

III. To evaluate the duration of response (DOR) and PFS in patients deriving clinical benefit (stable disease [SD], PR, CR) who continue therapy for an additional 12 months (24 total months).

CORRELATIVE OBJECTIVES:

I. To evaluate the changes in systemic immune activation, exhaustion, and T cell phenotypes in patients before and during treatment, and to compare these activation profiles between responding and progressing patients.

II. To profile the tumor microenvironment pre-treatment and monitor T cell dynamics and T-cell receptor (TCR) clonality by single-cell approaches before and during treatment, and compare these profiles between responding and progressing patients.

III. To determine lymphoma mutational profiles in peripheral blood circulating tumor DNA (ctDNA) and to compare changes in ctDNA levels and mutational profiling between responding and progressing patients.

IV. To evaluate DNA methylation (cytosine hydroxymethylation and cytosine methylation) status in cell free (cf)DNA at global level and to compare changes in cfDNA DNA methylation levels between responding and progressing patients.

OUTLINE:

Patients receive decitabine and cedazuridine orally (PO) once daily (QD) on days 1-3 or 1-5 of each cycle and nivolumab intravenously (IV) over 30 minutes on day 15 of each cycle. Treatment repeats every 28 days for 12 cycles in the absence of disease progression or unacceptable toxicity. Patients with CR, PR, or SD after 12 cycles receive decitabine and cedazuridine for an additional 12 months. Patients also undergo positron emission tomography (PET)/computed tomography (CT) and collection of blood samples throughout the trial.

After completion of study treatment, patients are followed up every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Dose Escalation: Histologically confirmed relapsed or refractory B cell lymphoma (non-Hodgkin lymphoma [NHL] or Hodgkin lymphoma [HL])
* Dose Expansion: Patients must have histologically confirmed relapsed or refractory DLBCL or HL
* Patients with DLBCL must have failed at least first line chemotherapy and must be transplant ineligible (either secondary to performance status or lack of adequate disease control or patient preference). Patients may be relapsed after autologous or allogeneic stem cell transplant (SCT), or after chimeric antigen receptor (CAR)-T cell therapy
* In dose escalation patients with HL or B cell NHL other than DLBCL must have relapsed after at least 2 lines of therapy and have no other curative options left. HL patients must be brentuximab vedotin refractory or intolerant. In dose expansion, patients with classic HL must have relapsed after at least 2 lines of therapy, and had autologous stem cell transplantation (ASCT), be ineligible for ASCT, or have refused ASCT. Prior treatment with checkpoint inhibitor is allowed
* Age >= 18 years. Because no dosing or adverse event data are currently available on the use of nivolumab in combination with ASTX727 in patients < 18 years of age, children are excluded from this study
* Eastern Cooperative Oncology Group (ECOG)/Karnofsky performance status =< 2 (Karnofsky >= 70%)
* Leukocytes >= 1,500/mcL (unless documented bone marrow involvement in which case lower values may be allowed)
* Absolute neutrophil count >= 1,000/mcL (unless documented bone marrow involvement in which case lower values may be allowed)
* Platelets >= 75,000/mcL (unless documented bone marrow involvement in which case lower values may be allowed)
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x institutional ULN
* Serum creatinine =< 1.5 x ULN OR creatinine clearance (CrCl) >= 50 mL/min (if using the Cockcroft-Gault formula)
* Patients with a requirement for steroid treatment or other immunosuppressive treatment: Patients should be excluded if they have a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression
* Patients with new or progressive brain metastases (active brain metastases) or leptomeningeal disease are eligible if the treating physician determines that immediate CNS specific treatment is not required and is unlikely to be required during the first cycle of therapy
* Patients with a prior malignancy that has completed treatment and or in remission for at least 3 years, or non-melanoma skin cancer or in situ cancer are eligible for this trial. Patients with concurrent malignancy or recent treatment for a concurrent malignancy are not eligible
* Patients should be New York Heart Association Functional Classification of class 2B or better
* The effects of nivolumab and ASTX727 on the developing human fetus are unknown. For this reason and because DNMTi agents as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential (WOCBP) and men must agree to use highly effective contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. WOCBP should use a highly effective contraception method to avoid pregnancy during treatment with ASTX727 and for at least 6 months after the last dose of investigational drug and must agree not to donate eggs (ova, oocytes) for the purpose of reproduction for the same time period. Women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]) within 24 hours prior to the start of nivolumab. An extension up to 72 hours prior to the start of study treatment is permissible in situations where results cannot be obtained within the standard 24-hour window. Women must not be breastfeeding. Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year. Men who are sexually active with WOCBP will be instructed to adhere to highly-effective contraceptive measures of birth control and not to father a child while receiving treatment and for a period of 3 months after the last dose of investigational product. Women who are not of childbearing potential (i.e., who are postmenopausal or surgically sterile as well as azoospermic men) do not require contraception

  * Women of childbearing potential (WOCBP) is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:
  * Women < 50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
  * Women ≥ 50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses > 1 year ago, had chemotherapy-induced menopause with last menses > 1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).

WOCBP receiving ASTX727 will be instructed to adhere to contraception for a period of 6 months after the last dose of investigational product. Men receiving ASTX727 and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 3 months after the last dose of investigational product. WOCBP receiving nivolumab as a single agent will be instructed to adhere to contraception for a period of 5 months after the last dose. These durations have been calculated using the upper limit of the half-life for nivolumab (25 days) and are based on the protocol requirement that WOCBP use contraception for 5 half-lives plus 30 days Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she (or the participating partner) should inform the treating physician immediately

* Ability to understand and the willingness to sign a written informed consent document. Participants with impaired decision-making capacity who have a legally-authorized representative (LAR) and/or family member available will also be eligible

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (2 weeks for Revlimid, 6 weeks for nitrosoureas or mitomycin C) prior to entering the study. Palliative (limited-field) radiation therapy is permitted, if all of the following criteria are met:

  * Repeat imaging demonstrates no new sites of bone metastases
  * The lesion being considered for palliative radiation is not a target lesion
* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1) with the exception of alopecia
* Patients who have had prior treatment with anti-PD-1/PD-L1 inhibitors or anti CTLA4 antibodies and were permanently discontinued from further treatment because of an adverse event. All other prior therapies are permissible. Prior checkpoint inhibitor therapy is allowed if there was no discontinuation due to adverse event
* Patients who are receiving any other investigational agents
* Patients with known brain metastases or leptomeningeal metastases may be excluded because of poor prognosis and concerns regarding progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ASTX727 or nivolumab, including severe hypersensitivity reaction to any monoclonal antibody
* Patients with uncontrolled intercurrent illness
* Patients with cognitive or other impairment that would prevent compliance with study requirements
* Pregnant women are excluded from this study because ASTX727 is a DNMTi agent and nivolumab is a PD-L1 inhibitor with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with ASTX727 and nivolumab, breastfeeding should be discontinued if the mother is treated with ASTX727 and nivolumab
* Patients with active autoimmune disease or history of autoimmune disease that might recur, which may affect vital organ function or require immune suppressive treatment including systemic corticosteroids, should be excluded. These include but are not limited to patients with a history of immune related neurologic disease, multiple sclerosis, autoimmune (demyelinating) neuropathy, Guillain-Barre syndrome (GBS), myasthenia gravis; systemic autoimmune disease such as systemic lupus erythematosus (SLE), connective tissue diseases, scleroderma, inflammatory bowel disease (IBD), Crohn's, ulcerative colitis, hepatitis; and patients with a history of toxic epidermal necrolysis (TEN), Stevens-Johnson syndrome, or phospholipid syndrome should be excluded because of the risk of recurrence or exacerbation of disease. Patients with vitiligo, endocrine deficiencies including thyroiditis managed with replacement hormones including physiologic corticosteroids are eligible. Patients with rheumatoid arthritis and other arthropathies, Sjogren's syndrome and psoriasis controlled with topical medication and patients with positive serology, such as antinuclear antibodies (ANA), anti-thyroid antibodies should be evaluated for the presence of target organ involvement and potential need for systemic treatment but should otherwise be eligible
* Patients who have had evidence of active or acute diverticulitis, intra-abdominal abscess, gastrointestinal (GI) obstruction and abdominal carcinomatosis which are known risk factors for bowel perforation should be evaluated for the potential need for additional treatment before coming on study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-11-03 (Actual); Primary Completion 2027-06-28 (Estimated); Study Completion 2027-06-28 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 2 years
  Frequency of subjects experiencing toxicities will be tabulated. Toxicities will be assessed and graded according to Common Terminology Criteria for Adverse Events version 5.0 terminology. Exact 95% confidence intervals around the toxicity proportions will be calculated.

SECONDARY OUTCOMES:
Complete response rate | Up to 2 years
  Will be reported along with the 95% confidence intervals.
Partial response rate | Up to 2 years
  Will be reported along with the 95% confidence intervals.
Overall response rate | Up to 2 years
  Will be reported along with the 95% confidence intervals.
Duration of response | Up to 2 years
  Will be estimated using Kaplan-Meier methodology. Greenwood's formula will be used to calculate 95% confidence intervals for the Kaplan-Meier estimates.
Overall survival | Up to 2 years
  Will be estimated using Kaplan-Meier methodology. Greenwood's formula will be used to calculate 95% confidence intervals for the Kaplan-Meier estimates.
Progression survival | Up to 2 years
  Will be estimated using Kaplan-Meier methodology. Greenwood's formula will be used to calculate 95% confidence intervals for the Kaplan-Meier estimates.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine S Diefenbach, Principal Investigator — Laura and Isaac Perlmutter Cancer Center at NYU Langone
Locations (9):
- United States (9):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Yale University, New Haven, Connecticut
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - NYU Langone Hospital - Long Island, Mineola, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm